CLINICAL TRIAL: NCT02472964
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group, Phase III Study of the Efficacy and Safety of Hercules Plus Taxane Versus Herceptin® Plus Taxane as First Line Therapy in Patients With HER2-Positive Metastatic Breast Cancer
Brief Title: Study of Efficacy and Safety of Myl1401O + Taxane vs Herceptin©+ Taxane for 1st Line, Met. Br. Ca.
Acronym: HERiTAge
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Mylan GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MYL-Her 3001; 2011-001965-42 (EudraCT Number)
Record Dates: First submitted 2015-06-03; First posted 2015-06-16 (Estimated); Results first posted 2018-10-30 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; hercules receptor kinase 2, Arabidopsis; Paclitaxel; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Herceptin© + Taxane (Active Comparator): Part 1: Herceptin© (trastuzumab) intravenously+ paclitaxel 80 mg/m2 weekly intravenously or docetaxel 75 mg/m2 intravenously once every three weeks (investigators choice) for 8 cycles then evaluate for primary endpoint.
  Part 2: If SD or PR, CR at cycle 9 (week 24) proceed to Herceptin© (trastuzumab) alone once every 3 weeks until DP or subject withdrawal .
  Interventions: Biological: Trastuzumab; Drug: Paclitaxel; Drug: Docetaxel
- MYL- 1401O + Taxane (Experimental): Part 1:MYL-1401O Intravenously + paclitaxel 80 mg/m2 weekly intravenously or docetaxel 75 mg/m2 intravenously once every three weeks (investigators choice) for 8 cycles then evaluate for primary endpoint.
  Part 2: If SD or PR, CR at cycle 9 (week 24) proceed to MYL-1401O alone once every 3 weeks until DP or subject withdrawal.
  Interventions: Biological: MYL- 1401O; Drug: Paclitaxel; Drug: Docetaxel

INTERVENTIONS:
Biological: Trastuzumab — Trastuzumab 8mg/kg Iv over 90 minutes x 1 then Trastuzumab 6 mg/kg IV over 30 minutes every 3 weeks
  Other Names: Herceptin©;
  Arms: Herceptin© + Taxane
Biological: MYL- 1401O — MYL-1401O 8mg/kg Iv over 90 minutes x 1 then HERMyl 1401O Trastuzumab 6 mg/kg IV over 30 minutes every 3 weeks
  Other Names: Hercules
  Arms: MYL- 1401O + Taxane
Drug: Paclitaxel — Paclitaxel 80mg/m2 IV over 60 minutes weekly.
Drug: Docetaxel — Docetaxel 75mg/m2 IV over 60 minutes on day 1 of a 3 week cycle

SUMMARY:
A multicenter, double-blind, randomized, parallel-group, Phase III study of the efficacy and safety of Hercules( Myl 1401O, Mylan Trastuzumab) plus taxane versus Herceptin® plus taxane as first line therapy in patients with HER2-positive metastatic breast cancer.

DETAILED DESCRIPTION:
Part 1: A multicenter, double-blind, randomized, parallel-group, Phase III study to compare the efficacy and safety of MYL-1401O (Mylan Trastuzumab biosimiliar) plus taxane versus Herceptin® plus taxane in patients with HER2+ MBC. Either docetaxel or paclitaxel (Investigator site level choice) is planned for at least 24 weeks until documented response to therapy, disease progression, or discontinuation. Disease response and progression will be assessed locally by the Investigator on the basis of clinical and radiographic evidence using RECIST 1.1 criteria. The primary and secondary efficacy analyses will be performed using independently assessed radiographic evidence for the Intent-to-Treat (ITT) population. The primary analysis population for best ORR will be those patients who had measureable disease at baseline and for the secondary endpoint, DR, only those who are responders will be included in the analysis.

Part 2: A multicenter, double-blind, parallel-group study to continue to compare the safety and immunogenicity and efficacy of MYL-1401O versus Herceptin® in patients with HER2+ MBC who have clinical benefit to first-line combination therapy with a taxane. All patients who have at least stable disease (SD), will continue with either single agent MYL-1401O or Herceptin® alone until death, unacceptable toxicity or disease progression.

Population pharmacokinetics: During Part 1 of the study, for both MYL-1401O, and Herceptin® treatment arms, PK sampling for Cmin and Cmax (end of infusion) will be collected for all patients. A PopPK subset, with sufficient samples available to perform the necessary analysis of PopPK modeling will be used to assess AUC, Cmax, Cmin, clearance, Vd, and T1/2 at various time points in the PopPK. Patients randomized into the main study will sign an additional consent form for the PopPK subset. We anticipate that approximately 80 patients will need to be enrolled in this subset collection in order to obtain sufficient samples for analysis.

Long term survival follow-up: OS for this treated population will be determined with every 3 month follow-up until either 240 deaths or 36 months, whichever occurs first, as observed from the time of randomization. The results for OS are expected to be reported March 2019. Exploratory evaluations: In addition, during Part 1 of the study, blood samples will be collected in all patients to assess the impact of soluble shed HER2/ECD on PK and efficacy at pre-dose on Cycles 1, 3, 5, 7, and end of treatment (EOT). Additional samples (ECD) will be obtained on Cycles 9, 13 and every 4 cycles thereafter, EOT and end of study (EOS) for continued evaluation of immunogenicity in patients continuing to receive therapy. A blood sample will be obtained on Cycle 1, Day 1, to be used for assay development and validation

ELIGIBILITY:
Inclusion Criteria:

Locally recurrent or MBC that is not amenable to curative surgery and/or radiation.

Documentation of HER2 gene amplification by fluorescent in situ hybridization (FISH) (as defined by a ratio >2.0) or documentation of HER2-overexpression by immunohistochemistry (IHC) (defined as IHC3+, or IHC2+ with FISH confirmation) based on the sponsor-identified central laboratory prior to randomization. Archival tumor tissue samples can be used.

Pathologically confirmed breast cancer with at least one measurable metastatic target lesion (based on RECIST criteria, version 1.1). Bone, central nervous system (CNS), and skin lesions, as well as lesions that were irradiated, biopsied or had any form of local intervention or surgical manipulation are only to be assessed as non-target lesions.

Patients previously treated with trastuzumab or lapatinib in the adjuvant setting are allowed if metastatic disease was diagnosed at least one year after the last dose of treatment.

Prior treatment with hormonal agents or bisphosphonates/denosumab is allowed. Bisphosphonates/denosumab can be given simultaneously with study treatment but cannot start after randomization and is considered an indication of progressive disease (PD). Hormonal agents must be discontinued prior to beginning study therapy.

Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 - 2

* Serum creatinine ≤1.5 x ULN (upper limit of normal),
* Total bilirubin ≤1.0 x ULN (>1.0 x ULN if documented Gilbert's disease),
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤2.5 x ULN,
* AST and/or ALT <1.5 x ULN if alkaline phosphatase >2.5 x ULN,
* Alkaline phosphatase >2.5 x ULN;if bone metastases present and no liver dysfunction present.

Left ventricular ejection fraction (LVEF) within institutional range of normal as measured by multiple gated acquisition scan or echocardiogram.

Exclusion Criteria:

Prior systemic therapy in the metastatic disease setting. This includes: chemotherapy, signal transduction inhibitors (e.g., lapatinib), HER2 targeted therapy (e.g., trastuzumab), or other investigational anticancer therapy.

Prior treatment with neoadjuvant or adjuvant anthracyclines with a cumulative dose of doxorubicin of >400 mg/m2, epirubicin dose >800 mg/m2.

Patients with bone or skin as the only site of disease. Patients with skin lesions measurable by CT scans or MRI as only site of measurable disease are allowed.

Surgery or radiotherapy ≤2 weeks preceding Day 1. Target lesions have to be outside the irradiated fields and the patient has fully recovered from surgery or radiotherapy.

Presence of unstable angina or a history of congestive heart failure according to the New York Heart Association criteria, history of myocardial infarction <1 year from randomization, clinically significant valvular disease, serious cardiac arrhythmia requiring treatment, uncontrolled hypertension or known pulmonary hypertension.

Peripheral sensory or motor neuropathy Grade 2 or higher according to the National Cancer Institute-Common Terminology Criteria (NCI-CTC) Version 4.03 [19].

Any other cancer, including contralateral breast cancer, within 5 years prior to screening with the exception of adequately treated ductal carcinoma in situ, adequately treated cervical carcinoma in situ, or adequately treated basal or squamous cell carcinoma of the skin.

Immunocompromized patients, including known seropositivity for human immunodeficiency virus, or current or chronic hepatitis B and/or hepatitis C infection (as detected by positive testing for hepatitis B surface antigen or antibody to hepatitis C virus with confirmatory testing).

Complete listing of Inc/Excl. within protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2012-07; Primary Completion 2016-03 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Pennella, MD, Study Director — Mylan Inc.
Locations (92):
- Brazil (12):
  - Mylan Investigational Site, Barretos
  - Mylan Investigational Site, Brasília
  - Mylan Investigational Site, Goiânia
  - Mylan Investigational Site, Ijuí
  - Mylan Investigational Site, Jaú
  - Mylan Investigational Site, Joinville
  - Mylan Investigational Site, Morumbi
  - Mylan Investigational Site, Porto Alegre
  - Mylan Investigational Site, Salvador
  - Mylan Investigational Site, Santo André
  - Mylan Investigational Site, São Paulo
  - Mylan Investigational Site, Sorocaba
- Chile (2):
  - Mylan Investigational Site, Santiago
  - Mylan Investigational Site, Temuco
- Georgia (2):
  - Mylan Investigational Site, Batumi
  - Mylan Investigational Site, Tbilisi
- Hungary (8):
  - Mylan Investigational Site, Budapest
  - Mylan Investigational Site, Debrecen
  - Mylan Investigational Site, Gyód
  - Mylan Investigational Site, Gyula
  - Mylan Investigational Site, Miskolc
  - Mylan Investigational Site, Nyíregyháza
  - Mylan Investigational Site, Szekszárd
  - Mylan Investigational Site, Szolnok
- India (13):
  - Mylan Investigational Site, Ahmedabad
  - Mylan Investigational Site, Bangalore
  - Mylan Investigational Site, Chennai
  - Mylan Investigational Site, Gūrgaon
  - Mylan Investigational Site, Hyderabad
  - Mylan Investigational Site, Jaipur
  - Mylan Investigational Site, Karamsad
  - Mylan Investigational Site, Madurai
  - Mylan Investigational Site, Mumbai
  - Mylan Investigational Site, Nashik
  - Mylan Investigational Site, Pune
  - Mylan Investigational Site, Surat
  - Mylan Investigational Site, Vijaywada
- Latvia (3):
  - Mylan Investigational Site, Daugavpils
  - Mylan Investigational Site, Leipaja
  - Mylan Investigational Site, Riga
- Peru (3):
  - Mylan Investigational Site, Arequipa
  - Mylan Investigational Site, Lima
  - Mylan Investigational Site, Surquillo
- Romania (9):
  - Mylan Investigational Site, Brasov
  - Mylan Investigational Site, Bucharest
  - Mylan Investigational Site, Cluj-Napoca
  - Mylan Investigational Site, Constanța
  - Mylan Investigational Site, Craiva
  - Mylan Investigational Site, Făurei
  - Mylan Investigational Site, Iași
  - Mylan Investigational Site, Oradea
  - Mylan Investigational Site, Timișoara
- Russia (9):
  - Mylan Investigational Site, Arkhangelsk
  - Mylan Investigational Site, Ivanovo
  - Mylan Investigational Site, Kazan'
  - Mylan Investigational Site, Kursk
  - Mylan Investigational Site, Moscow
  - Mylan Investigational Site, Rostov-on-Don
  - Mylan Investigational Site, Ryazan
  - Mylan Investigational Site, Saint Petersburg
  - Mylan Investigational Site, Samara
- Serbia (3):
  - Mylan Investigational Site, Belgrade
  - Mylan Investigational Site, Kamenica
  - Mylan Investigational Site, Sremska
- Slovakia (4):
  - Mylan Investigational Site, Bardejov
  - Mylan Investigational Site, Košice
  - Mylan Investigational Site, Nové Zámky
  - Mylan Investigational Site, Trnava
- South Africa (8):
  - Mylan Investigator Site, Bloemfontein
  - Mylan Investigator Site, Durban
  - Mylan Investigational Site, George
  - Mylan Investigational Site, Johannesburg
  - Mylan Investigator Site, Kraaifontein
  - Mylan Investigational Site, Port Elizabeth
  - Mylan Investigational Site, Pretoria
  - Mylan Investigational Site, Vereeniging
- Thailand (5):
  - Mylan Investigator Site, Bangkok
  - Mylan Investigator Site, Chiang Mai
  - Mylan Investigator Site, Phitsanulok
  - Mylan Investigator Site, Rajthavee
  - Mylan Investigator Site, Songkhla
- Turkey (Türkiye) (4):
  - Mylan Investigator Site, Ankara
  - Mylan Investigator Site, Istanbul
  - Mylan Investigator Site, Izmir
  - Mylan Investigator Site, Kocaeli
- Ukraine (7):
  - Mylan Investigator Site, Cherkassy
  - Mylan Investigator Site, Chernivtsi
  - Mylan Investigator Site, Dnipropetrovsk
  - Mylan Investigator Site, Lutsk
  - Mylan Investigator Site, Lviv
  - Mylan Investigator Site, Sumy
  - Mylan Investigator Site, Uzhhorod

REFERENCES:
- [Derived] Rugo HS, Pennella EJ, Gopalakrishnan U, Hernandez-Bronchud M, Herson J, Koch HF, Loganathan S, Deodhar S, Marwah A, Manikhas A, Bondarenko I, Mukhametshina G, Nemsadze G, Parra JD, Abesamis-Tiambeng MLT, Baramidze K, Akewanlop C, Vynnychenko I, Sriuranpong V, Mamillapalli G, Roy S, Yanez Ruiz EP, Barve A, Fuentes-Alburo A, Waller CF. Final overall survival analysis of the phase 3 HERITAGE study demonstrates equivalence of trastuzumab-dkst to trastuzumab in HER2-positive metastatic breast cancer. Breast Cancer Res Treat. 2021 Jul;188(2):369-377. doi: 10.1007/s10549-021-06197-5. Epub 2021 Jun 14. PMID 34125340
- [Derived] Rugo HS, Barve A, Waller CF, Hernandez-Bronchud M, Herson J, Yuan J, Sharma R, Baczkowski M, Kothekar M, Loganathan S, Manikhas A, Bondarenko I, Mukhametshina G, Nemsadze G, Parra JD, Abesamis-Tiambeng ML, Baramidze K, Akewanlop C, Vynnychenko I, Sriuranpong V, Mamillapalli G, Ray S, Yanez Ruiz EP, Pennella E; Heritage Study Investigators. Effect of a Proposed Trastuzumab Biosimilar Compared With Trastuzumab on Overall Response Rate in Patients With ERBB2 (HER2)-Positive Metastatic Breast Cancer: A Randomized Clinical Trial. JAMA. 2017 Jan 3;317(1):37-47. doi: 10.1001/jama.2016.18305. PMID 27918780

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 500 subjects enrolled at 95 sites across Eastern Europe, Russia, Asia Pacific, Africa and South America. The intent to treat1(ITT1) population of 458 was used to determine Primary Outcome of Overall Response Rate.
Pre-assignment Details: The primary efficacy analysis was derived fromITT1 population 230 (MYL-1401O) + 228 (Herceptin)= 458. Safety analysis was derived from the Safety Population 247(MYL-1401O)+246(Herceptin)= 493. Total Randomized population 249(MYL-1401O) +251(Herceptin)= 500.
Groups:
- HerMyl 1401O Trastuzumab + Taxane: Part 1:Myl 1401OTrastuzumab Intravenously + paclitaxel 80 mg/m2 weekly intravenously or docetaxel 75 mg/m2 intravenously once every three weeks (investigators choice) for 8 cycles then evaluate for primary endpoint.
  Part 2: If SD or PR, CR at cycle 9 (week 24) proceed to Myl 1401O( Mylan Trastuzumab) alone once every 3 weeks until DP or subject withdrawal.
Period: Part 1 (up to Week 24)
Arm/Group | Herceptin© + Taxane | HerMyl 1401O Trastuzumab + Taxane
Started (The disposition of the patients has been provided for the safety sample population.) | 246 | 247
Completed | 171 | 185
Not Completed | 75 | 62
Not completed — Adverse Event | 2 | 4
Not completed — disease progression | 58 | 47
Not completed — Death | 3 | 6
Not completed — Physician Decision | 3 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 7 | 2
Not completed — Other | 2 | 1
Period: Part 2 (Week 24-week 48)
Arm/Group | Herceptin© + Taxane | HerMyl 1401O Trastuzumab + Taxane
Started (The disposition of the patients has been provided for the safety sample.) | 163 | 179
Completed | 98 | 116
Not Completed | 65 | 63
Not completed — Adverse Event | 4 | 2
Not completed — Disease Progression | 52 | 56
Not completed — Death | 0 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Protocol Violation | 3 | 1

BASELINE CHARACTERISTICS:
Population: Bseline Analysis Population Description: The primary efficacy endpoint analysis was conducted in the intention to treat (IIT)population ( only those patients randomized after the second amendment of the protocol)
Groups:
- Herceptin© + Taxane: Part 1: Herceptin© (trastuzumab) intravenously+ paclitaxel 80 mg/m2 weekly intravenously or docetaxel 75 mg/m2 intravenously once every three weeks (investigators choice) for 8 cycles then evaluate for primary endpoint.
  Part 2: If SD or PR, CR at cycle 9 (week 24) proceed to Herceptin© (trastuzumab) alone once every 3 weeks until DP or subject withdrawal .
  Herceptin© 8mg/kg Iv over 90 minutes x 1 then Herceptin© 6 mg/kg IV over 30 minutes every 3 weeks
  Paclitaxel 80mg/m2 IV over 60 minutes weekly.
  Docetaxel 75mg/m2 IV over 60 minutes on day 1 of a 3 week cycle
- MYL-1401O + Taxane: Part 1:MYL-1401O intravenously + paclitaxel 80 mg/m2 weekly intravenously or docetaxel 75 mg/m2 intravenously once every three weeks (investigators choice) for 8 cycles then evaluate for primary endpoint.
  Part 2: If SD or PR, CR at cycle 9 (week 24) proceed to Myl 1401O alone once every 3 weeks until DP or subject withdrawal.
  MYL-1401O 8mg/kg Iv over 90 minutes x 1 then MYL-1401O 6 mg/kg IV over 30 minutes every 3 weeks
  Paclitaxel 80mg/m2 IV over 60 minutes weekly.
  Docetaxel 75mg/m2 IV over 60 minutes on day 1 of a 3 week cycle
- Total: Total of all reporting groups
Arm/Group | Herceptin© + Taxane | MYL-1401O + Taxane | Total
Number analyzed (Participants) | 228 | 230 | 458
Age, Customized [Count of Participants; unit: Participants] — Population: The primary efficacy endpoint analysis was conducted in the intention to treat (IIT1)population ( only those patients randomized after the second amendment of the protocol)
  Participants
    < 50years of age | 86 | 74 | 160
    >/= 50years of age | 142 | 156 | 298
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 228 | 230 | 458
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The primary efficacy endpoint analysis was conducted in the intention to treat (IIT1)population ( only those patients randomized after the second amendment of the protocol)
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 72 | 70 | 142
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 1 | 3
    White | 154 | 159 | 313
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Chile | 4 | 1 | 5
  Czechia | 1 | 0 | 1
  Georgia | 23 | 26 | 49
  Hungary | 8 | 5 | 13
  India | 31 | 24 | 55
  Latvia | 2 | 4 | 6
  Philippines | 18 | 30 | 48
  Poland | 6 | 13 | 19
  Romania | 5 | 3 | 8
  Russia | 73 | 71 | 144
  Serbia | 2 | 3 | 5
  Slovakia | 1 | 2 | 3
  South Africa | 3 | 8 | 11
  Thailand | 23 | 16 | 39
  Ukraine | 28 | 24 | 52

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint : Compare Best Overall Response Rate (ORR) (According to Response Evaluation Criteria in Solid Tumor [RECIST] 1.1 Criteria) at Week 24 of MYL-1401O Plus Taxane Versus Herceptin® Plus Taxane in the ITT1 Population
Description: Tumor measurements were perform by centralized blinded reviewers using RECIST 1.1 criteria. Per RECIST 1.1: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph node must have reduction in short axis to <10 mm.Partial Response (PR): >/= 30% decrease sum of the diameters of target lesions from baseline sum diameters.
  Progressive Disease (PD): </= 20% increase in the sum of the diameters of target lesions, from the smallest sum on study with at least a 5 mm absolute increase in the sum of all lesions. The appearance of one or more new lesions* denotes disease progression.
  Stable Disease (SD): Neither sufficient decrease or increase. Evaluation of Non-Target Lesions Complete Response (CR): Disappearance of all non-target lesions. Non-complete Response/Non-Progressive Disease: Persistence of one or more non-target lesions. Progressive Disease (PD): Substantial, unequivocal progression of existing non-target lesions.
Time Frame: from time of First treatment to week 24
Population: The primary efficacy analysis was conducted in the Intent To Treat population 1 (ITT1) ( all patients randomized after Amendment 2 of the protocol)
Measure: Count of Participants; unit: Participants
Groups:
- MYL-1401O Trastuzumab + Taxane: Part 1:Myl 1401OTrastuzumab Intravenously + paclitaxel 80 mg/m2 weekly intravenously or docetaxel 75 mg/m2 intravenously once every three weeks (investigators choice) for 8 cycles then evaluate for primary endpoint.
  Part 2: If SD or PR, CR at cycle 9 (week 24) proceed to Myl 1401O( Mylan Trastuzumab) alone once every 3 weeks until DP or subject withdrawal.
Arm/Group | Herceptin© + Taxane | MYL-1401O Trastuzumab + Taxane
Number analyzed (Participants) | 228 | 230
Participants
  Complete Response | 0 | 3
  Partial Response | 146 | 157
  Stable Disease | 49 | 48
  Progressive Disease | 20 | 9
  Not Evaluable | 13 | 13

ADVERSE EVENTS:
Time Frame: ICF until 28 days( +/- 7 days) after last dose of IMP per patient. The active reporting period for AEs is from the time the patient receives the first dose until 28 days( +/- 7 days) after last administered dose of IMP per patient. However, SAEs should be reported any time after the active reporting period, when the Investigator becomes aware and the SAE is considered to be reasonably related to the study drug.
Description: The Investigator is responsible for the detection and documentation of events meeting the criteria and definition of an AE or SAE, as described previously. At each visit, the patient will be allowed time to spontaneously report any issues since the last visit or evaluation.
  The Investigator will then monitor and/or ask about or evaluate AEs using non-leading questions. Any clinically relevant observations made during the visit are also to be considered AEs.
Groups:
- Myl 1401O Trastuzumab + Taxane: Part 1:Myl 1401OTrastuzumab Intravenously + paclitaxel 80 mg/m2 weekly intravenously or docetaxel 75 mg/m2 intravenously once every three weeks (investigators choice) for 8 cycles then evaluate for primary endpoint.
  Part 2: If SD or PR, CR at cycle 9 (week 24) proceed to Myl 1401O( Mylan Trastuzumab) alone once every 3 weeks until DP or subject withdrawal.
Arm/Group | Herceptin© + Taxane | Myl 1401O Trastuzumab + Taxane
Serious Adverse Events (participants affected / at risk) | 91/246 | 97/247
Other Adverse Events (participants affected / at risk) | 232/246 | 229/247
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Herceptin© + Taxane (N=246) | Myl 1401O Trastuzumab + Taxane (N=247)
Febrile Neutropenia (Blood and lymphatic system disorders) | 10 | 11
Leukopenia (Blood and lymphatic system disorders) | 12 | 5
Neutropenia (Blood and lymphatic system disorders) | 62 | 68
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 2
Carditis (Cardiac disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Anal Fissure (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 3
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Toxicity (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Rectal Perforation (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
Death (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Hyperthermia (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Multi-Organ Failure (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 1 | 1
Anaphylactic Reaction (Immune system disorders) | 0 | 2
Drug Hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 0
Bronchitis (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 3
Influenza (Infections and infestations) | 1 | 0
Mastitis (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 6
Rectal Abscess (Infections and infestations) | 1 | 0
Renal Abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 0
Septic Shock (Infections and infestations) | 0 | 1
Tubo-Ovarian Abscess (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 2
Wound Infection (Infections and infestations) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 | 0
Blood Uric Acid Increased (Investigations) | 1 | 1
Ejection Fraction Decreased (Investigations) | 0 | 1
White Blood Cell Count Decreased (Investigations) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 1 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Lymphanangiosis Carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Accelerated Hypertension (Vascular disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Peripheral Ischaemia (Vascular disorders) | 0 | 1
Thrombophlebitis Superficial (Vascular disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Herceptin© + Taxane (N=246) | Myl 1401O Trastuzumab + Taxane (N=247)
Alopecia (Skin and subcutaneous tissue disorders) | 135 | 143
Neutropenia (Blood and lymphatic system disorders) | 83 | 91
Neuropathy Peripheral (Nervous system disorders) | 30 | 31
Diarrhea (Gastrointestinal disorders) | 49 | 50
Asthenia (Musculoskeletal and connective tissue disorders) | 41 | 57
Leukopenia (Blood and lymphatic system disorders) | 42 | 40
Nausea (Gastrointestinal disorders) | 37 | 51
Anemia (Blood and lymphatic system disorders) | 44 | 41
Oedema Peripheral (General disorders) | 31 | 38
Fatigue (General disorders) | 36 | 30
Pyrexia (General disorders) | 31 | 24
Myalgia (Musculoskeletal and connective tissue disorders) | 23 | 25
Vomiting (Gastrointestinal disorders) | 21 | 26
Decreased Appetite (Gastrointestinal disorders) | 25 | 23
Rash (Skin and subcutaneous tissue disorders) | 25 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 33
Alanine Aminotransferase Increased (Investigations) | 22 | 22
Urninary Tract Infection (Infections and infestations) | 18 | 23
Nail Disorder (Skin and subcutaneous tissue disorders) | 22 | 17
Aspartate Amniotransferase Increased (Investigations) | 24 | 16
Hyperglycemia (Metabolism and nutrition disorders) | 19 | 15
Bone Pain (Musculoskeletal and connective tissue disorders) | 14 | 21
Headache (Nervous system disorders) | 28 | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 19
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 | 15
Infusion Related Reaction (Injury, poisoning and procedural complications) | 11 | 17
Peripheral Sensory Neuropathy (Nervous system disorders) | 36 | 32
Peripheral Swelling (General disorders) | 13 | 11
Upper Respiratory Infection (Infections and infestations) | 5 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes